CLINICAL TRIAL: NCT00220506
Title: Fatigue Treatment Using Provigil in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Fatigue Treatment Using Provigil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3769-MD-CTIL
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-02-17 (Estimated); Status verified 2006-02

CONDITIONS: All Multiple Sclerosis Patients
Keywords: provigil; fatigue; Multiple Sclerosis; cognition
MeSH Terms: conditions — Fatigue; Multiple Sclerosis | interventions — Modafinil

INTERVENTIONS:
Drug: Provigil

SUMMARY:
To determine whether therapy with Modafinal(Provigil) is safe and effective in fatigue in MS Patients

DETAILED DESCRIPTION:
Multiple sclerosis and fatigue Fatigue is one of the most common symptoms of multiple sclerosis (MS), occurring in 30%-80% of patients and for many of them fatigue is the most disabling symptom (1).

Definition of fatigue according to the MS Council for Clinical Practice Guidelines is as follows: "A subjective lack of physical and/or mental energy that is perceived by the individual or caregiver to interfere with usual and desired activities".

As fatigue is a subjective and non-specific symptom, and can easily be confused with either weakness or depressed mood, both common in MS, the following characteristics have been defined to better diagnose MS-associated fatigue:

* MS-related fatigue generally occurs on a daily basis.
* It tends to worsen as the day progresses.
* It tends to be aggravated by heat and humidity.
* It is not directly correlated with either depression or the degree of physical impairment.
* It may occur first thing in the morning even if the patient has had a restful full night's sleep.

The current medications used for the treatment of MS-associated fatigue such as amantadine hydrochloride and pemoline are useful to some, but not all patients. In a multicenter trial (2) it was found that 100 mg amantadine twice daily significantly improves fatigue. Pemoline in a placebo-controlled trial (3) failed to show significant effect on fatigue in MS patients and was poorly tolerated as side effects occurred in 25% of patients. A third trial (4) compared pemoline to amantadine and placebo, and showed only a positive trend for pemoline, while amantadine had a benefit over placebo in some fatigue measures. There was also a marked placebo effect in this trial, with approximately half of patients reporting improvement in fatigue no matter what treatment (pemoline, amantadine or placebo) they were taking.

In the current study proposal we intend to evaluate the effect of Provigil on MS-associated fatigue.

The possibility for add-on drug that will affect fatigue in MS is of importance, as fatigue has a significant impact on activities of daily living, interfering with work, family life and social activities.

1.2. The fatigue scale named "Fatigue Impact Scale" The awareness of the impact of fatigue on patient's quality of life (QOL) and the need to evaluate the effect of the different therapies on this parameter resulted in the development and validation of different questionnaires for the measurement of fatigue, i.e., the Fatigue Impact Scale (FIS), which has been shown to measure both, fatigue and treatment effect on fatigue (6-9).

The FIS is a reliable and validated 40-items questionnaire that is capable of selecting a treatment effect. It is a made up of 3 sub-scales: physical, cognitive and social. Each question is scored from 0-4, allowing a total score of 160. High scores indicate high impairment.

ELIGIBILITY:
Inclusion Criteria:

* The patients should be diagnosed with clinically definite MS (Posner criteria).
* EDSS at screening: 0 to 5.5, inclusive.
* Positive Fatigue impact scale 40 points or more.
* Age 18-55 years.
* Co-operating patient, capable of complying with all of trial procedures (i.e. FIS, QOL, etc…).
* Patient who signed written informed consent.
* Women of childbearing potential must use effective birth control method during study.

Exclusion Criteria:

* Life threatening and/or unstable clinical condition which in the opinion of the investigator might compromise trial completion
* A relapse during the last 30 days prior to the study.
* Systemic steroid therapy within 30 days
* Known hypersensitivity or intolerance, to Provigil or related substances or to any component of the formulation.
* Sleep apnea
* Narcolepsy
* Participation in experimental drug trials during the last 30 days prior to the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2005-09; Study Completion 2006-12

PRIMARY OUTCOMES:
To determine fatigue impact scale

SECONDARY OUTCOMES:
to determine cognition measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dolev, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Multiple Sclerosis Center, Tel Litwinsky, Israel